CLINICAL TRIAL: NCT00535457
Title: The Effects of Pre-operative Magic Tricks Performance on Pre-operative Anxiety in Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ze'ev Shenkman, MD, Sheba Medical Center, Department of Anesthesia C
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHEBA-07-4786-ZS-CTIL
Record Dates: First submitted 2007-09-23; First posted 2007-09-26 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Anxiety
Keywords: anxiety; maladaptive behavior; anesthesia; Anxiety before anesthesia and maladaptive behavior after anesthesia.
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Children will watch tricks ("magic") before anesthesia induction
  Interventions: Other: Preoperative Magic Tricks

INTERVENTIONS:
Other: Preoperative Magic Tricks — Watching "magic"; Study patients will watch the anesthesiologist performing tricks ("magic") before anesthesia induction.

SUMMARY:
It is not uncommon for children to undergo surgery. Surgery is a threatening event that is composed of various stress-provoking stimuli. Pre-operative anxiety is a common emotional response among operated children and their parents. In the current study we are going to examine if tricks done by the anesthesiologist before anesthetic induction are equally as effective as oral midazolam premedication in the reduction of pre-operative anxiety in children before and after surgery. A successful anxiety reduction may be advantageous over pharmacological premedication by cost reduction, a possibly shorter post anesthesia care stay and by reducing postoperative maladaptive behavior rate.

Study hypothesis: 1. similar anxiety scores will be observed in children that will watch their anesthesiologist performing tricks and in those who will receive oral midazolam premedication but no tricks.

2. Similar rates of postoperative maladaptive behavior will be found in children that that will see tricks and in those that will receive midazolam premedication.

ELIGIBILITY:
Inclusion Criteria:

* age 3-12 years
* minor surgeries / diagnostic procedures such as endoscopy, biopsy

Exclusion Criteria:

* children that do not speak Hebrew
* American Society of Anesthesiologists (ASA) status above II
* a need for regional anesthesia only
* a need for an intravenous (IV) cannulation at the induction room or operating room before the induction of anesthesia.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
anxiety scores | Technical problems with video-taping of the patients still avoid us from recruiting patients. Therefore, the time frame of the study is still unclear tome.
postoperative maladaptive behavior rate

SECONDARY OUTCOMES:
preoperative anxiety scores and rate of postoperative maladaptive behavior

CONTACTS AND LOCATIONS:
Overall Officials: Ze'ev Shenkman, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel